CLINICAL TRIAL: NCT05424705
Title: Prediction of Atherosclerotic Plaque Progression in Patients With Acute Coronary Syndrome
Brief Title: Prediction of Atherosclerotic Plaque Progression
Acronym: PPP
Status: Active, not recruiting | Type: Observational
Sponsor: Na Homolce Hospital (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: Principal Investigator, Karel Kopriva, M.D, Na Homolce Hospital
Other Study IDs: 140504
Record Dates: First submitted 2022-05-16; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient DNA will be isolated from peripheral blood leucocytes by standard techniques. Genetic analysis of polymorphisms in gene for Hemoxygenase-1 and endothelial Nitric Oxide Synthase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OCT, NIRS

SUMMARY:
To predict coronary atherosclerosis progression in patients with acute coronary syndrome by the use of intracoronary imaging methods.

To investigate the ability of NIRS to detect vulnerable plaque characterized by the presence of OCT-defined TCFA To study the influence of gene polymorphisms (in genes playing role in vessel dilatation) on the progression of coronary atherosclerosis and clinical outcomes

DETAILED DESCRIPTION:
The fundamental aim of this study is to investigate the ability of intracoronary imaging to predict progression of coronary atherosclerosis in patients with acute coronary syndrome. In patients who are indicated for acute coronary angiography and have at least one non-culprit lesion (not indicated for revascularization) identical segment of non-culprit vessel will be analysed and several parameters will be detected by OCT (optical coherence tomography) and NIRS (near-infrared spectroscopy) including the presence of TCFA (thin-cap fibroatheroma) and plaque lipid content quantified by LCBI (lipid core burden index). During follow up visits (1Y, 2Y, 5Y and 10Y) major cardiovascular events will be monitored and the progression of coronary involvement will be estimated at 1Y and 2Y by CCTA (coronary computed angiography).

The second part of the trial is to investigate the ability of NIRS to detect vulnerable plaque characterized by the presence of OCT-defined TCFA.

A further target is to study the influence of gene polymorphisms (in genes playing a role in vessel dilatation) on the progression of coronary atherosclerosis and clinical outcomes. Patient DNA will be isolated from peripheral blood leucocytes, and polymorphisms in genes for Hemoxygenase-1 and endothelial Nitric Oxide Synthase will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome diagnosis
* Presence of at least one non-culprit coronary lesion (not indicated for revascularisation)

Exclusion Criteria:

* Contraindication for OCT or IVUS
* Circulatory instability
* Renal insufficiency (creatinine level >200umol/l)
* Pregnant or of childbirth age and not using reliable contraception
* Life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome indicated for coronary angiography with presence of a non-culprit lesion not indicated for revascularization
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of coronary atherosclerosis progression | Two years from the date of cardiac catheterization
  Prediction of coronary atherosclerosis progression (assesed by computed tomography, CT) in patients with acute coronary syndrome by the use of intracoronary imaging methods (OCT and NIRS)

SECONDARY OUTCOMES:
Detection of vulnerable coronary atherosclerotic plaques by NIRS and OCT | Measured once at the time of cardiac catheterization.
  Subjects are presenting for their clinically-indicated cardiac catheterization and NIRS and OCT imaging are performed at the time of this catheterization).
  NIRS is used for the quantification of plaque lipid content using the 4mm region of the vessel with the highest lipid core burden index (LCBI) and thus, the highest lipid content (maxLCBI4mm). OCT is used for the measuring of the thickness of plaque fibrous cap and thus, the presence of thin-cap fibroatheroma (TCFA).
Presence of gene polymorphisms | Analyzed once at the time of cardiac catheterization.
  Presence of gene polymorphisms in genes for Hemoxygenase-1 ane Endothelial Nitric Oxide Synthase by genetic analysis of patient DNA isolated from periferal blood leukocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided